CLINICAL TRIAL: NCT04812717
Title: Prevention of Vasoplegia With the Use of CytoSorb.
Brief Title: Prevention of Low Blood Pressure After Cardiac Surgery in Heart Failure Patients With a Filter Called CytoSorb.
Acronym: CytoSorb-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meindert Palmen, MD PhD, Cardiothoracic Surgeon, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P20.039; NL71623.058.20 (Other: Central Committee on Research Involving Human Subjects(CCMO))
Record Dates: First submitted 2021-03-16; First posted 2021-03-24 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure; Vasoplegia
Keywords: Heat Failure; Vasoplegia; Cardiopulmonary Bypass; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Heart Failure; Vasoplegia; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Perfusionists will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CytoSorb-Yes (Active Comparator): Heart failure patients that will receive intraoperative treatment with CytoSorb.
  Interventions: Device: CytoSorb device
- CytoSorb-No (No Intervention): Heart failure patients that will not receive intraoperative treatment with CytoSorb.

INTERVENTIONS:
Device: CytoSorb device — The CytoSorb device will be placed in the CPB circuit in half of the study population during their cardiac operation.
  Arms: CytoSorb-Yes

SUMMARY:
Vasoplegia is a common complication after heart surgery for heart failure. With vasoplegia, the blood vessels can no longer squeeze properly, causing low blood pressure that is sometimes difficult to treat with medication. One of the causes of this complication is likely to be the use of the heart-lung machine, a device that takes over the function of the heart and lungs during surgery. The blood then comes into contact with a foreign environment and this can cause a reaction of the immune system. Patients with heart failure are extra sensitive to this reaction.

CytoSorb device is a filter that can be built into the heart-lung machine and can reduce the response of the immune system. Therefore, this study aims to investigate whether the use of this filter during heart surgery in patients with heart failure results in a less frequent occurrence of vasoplegia after surgery.

DETAILED DESCRIPTION:
The incidence and prevalence of chronic heart failure is increasing. Despite the expansion of therapeutic options, overall survival and quality-of-life remain poor. When optimal medical therapy and cardiological interventions have failed to improve a patient's condition, surgical intervention may be a valid option in order to improve cardiac function. Different surgical treatments have improved clinical outcome. Unfortunately, heart failure surgery is associated with an increased risk of vasoplegia. This syndrome is characterized by hypotension and the continuous need of vasopressors, despite a normal or high cardiac index. The incidence of vasoplegia ranges from 11-31% in patients undergoing heart failure surgery. The prognosis of vasoplegia is poor. Prolonged hypotension and the accompanying hypoperfusion lead to end-organ dysfunction and is associated with an increased morbidity and mortality. The investigators hypothesise that the balance of the vascular system of patients with heart failure is fragile and therefore could easily be disturbed by a systemic inflammatory response syndrome (SIRS) caused by the cardiopulmonary bypass (CPB) and surgical trauma, making these patients more prone to develop vasoplegia. Minimising this SIRS reaction could be a strategy to prevent vasoplegia. Therefore, the objective of this single-center, investigator-initiated study is to analyse the efficacy and cost-effectiveness of using CytoSorb in preventing vasoplegia in patients with heart failure undergoing cardiac surgery on CPB.

CytoSorb treatment will be conducted intraoperatively and the device will be applied in a parallel circuit in the CPB. The total study intervention protocol takes 5 days and starts on the day of the surgery (day 0) and ends at day 4 postoperatively. Patient clinical data will be collected until day 30.

The vascular reactivity in response to a vasoconstrictor will be assessed in all patients at 3 different time points (after induction, after CPB, on day 1 postoperatively). During the vasoconstriction test, a bolus of 2 μg/kg phenylephrine is administered intravenously, after which the effect on the systemic vascular resistance is registered. At the same time points and in addition, before induction (baseline) and on day 4 the sublingual microcirculation will be monitored and blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HF in line with the European Society of Cardiology (ESC) guidelines34;
* Left ventricular EF ≤35%;
* Undergoing cardiac surgery on CPB with an anticipated duration of >120 minutes;
* Age ≥18 years.

Exclusion Criteria:

* Incapacitated;
* Emergency operation;
* Need for moderate or high dosages of intravenous inotropic support (>4 gamma dobutamine or dopamine) and/or vasopression;
* Severe tricuspid regurgitation;
* Daily use of nitroglycerine or isosorbide dinitrate;
* Use of alpha blockers;
* Being heparin-induced thrombocytopenia (HIT) positive and citrate regional anticoagulation is unavailable as an alternative anticoagulation method;
* Platelet count <20,000/μL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Delta systemic vascular resistance index (SVRi) after CPB. | during surgery (2-10 hours)
  The change in SVRi after the administration of phenylephrine after cessation of CPB.
Incidence of vasoplegia. | 72 hours
  Vasoplegic syndrome defined as the continuous need of vasopressors (norepinephrine ≥0.2 μg/kg/min for at least 12 consecutive hours, terlipressin, or methylene blue) in combination with a cardiac index (CI) ≥2.2 l/min/m2 for at least 12 consecutive hours, starting within the first 3 days postoperatively.

SECONDARY OUTCOMES:
Delta SVRi in ICU. | postoperative day 1
  The change in SVR after the administration of phenylephrine during the postoperative day one in the Intensive Care Unit (ICU).
Total administered dosage of vasopressors. | 30 days
Change in IL-6, IL-8, IL-10 levels. | until postoperative day 4 (96 hours)
Change in microvascular flow index [MFI],heterogeneity index [HI]. | until postoperative day 4 (96 hours)
  Heterogeneity index [HI] will be calculated as the difference between the highest MFI minus the lowest MFI and divided by the mean MFI.
Change in capillary density, functional capillary density [FCD], total vessel density [TVD], perfused vessel density [PVD]. | until postoperative day 4 (96 hours)
Change in proportion of perfused vessels [PPV]. | until postoperative day 4 (96 hours)
Change in rolling leucocytes [RL] levels. | until postoperative day 4 (96 hours)
Change in mean cell velocity [MCV], red blood cell velocity [RBCv]. | until postoperative day 4 (96 hours)
Change in capillary hematocrit. | until postoperative day 4 (96 hours)
Change in mean arterial pressure (MAP) after phenylephrine administration. | until postoperative day 1 (24 hours)
Hours on mechanical ventilation. | 30 days
Hours on mechanical circulatory support. | 30 days
Hours on postoperative renal replacement therapy. | 30 days
End organ damage (kidney dysfunction). | 30 days
Change in total Sequential Organ Failure Assessment Score (SOFA). | 30 days
Amount of used resuscitation fluids. | 30 days
Amount of used blood transfusion products. | 30 days
Length of ICU stay. | 30 days
Length of hospital stay. | 30 days
30-Day hospital readmissions. | 30 days
All-cause mortality. | 30 days

OTHER OUTCOMES:
Costs. | 30 days
  Market prices will be used for the CytoSorb intervention, vasopressor and inotropic medication, amount of blood transfusion products and resuscitation fluids, and reference prices from the Dutch guidelines for economic evaluations in healthcare for duration of surgery, ICU stay, and non-ICU hospital stay, hospital readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Meindert Palmen, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Papazisi O, Bruggemans EF, Berendsen RR, Hugo JDV, Lindeman JHN, Beeres SLMA, Arbous MS, van den Hout WB, Mertens BJA, Ince C, Klautz RJM, Palmen M. Prevention of vasoplegia with CytoSorb in heart failure patients undergoing cardiac surgery (CytoSorb-HF trial): protocol for a randomised controlled trial. BMJ Open. 2022 Sep 19;12(9):e061337. doi: 10.1136/bmjopen-2022-061337. PMID 36123067